CLINICAL TRIAL: NCT05800470
Title: The Novel Application of fNIRS-based Neurofeedback to Enhance Effects of Motor Imagery on Balance and Gait Performance in Individuals With Parkinson's Disease
Brief Title: The Effects of fNIRS-based Neurofeedback Training on Balance and Gait in Parkinson's Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Principal Investigator, Ray-Yau Wang, Professor, National Yang Ming Chiao Tung University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: NYCU112020AE
Record Dates: First submitted 2023-02-22; First posted 2023-04-05 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Parkinson Disease; Movement Disorder, Functional
Keywords: Neurofeedback; Motor imagery; Parkinson's disease
MeSH Terms: conditions — Parkinson Disease; Conversion Disorder

STUDY DESIGN:
Intervention Model Description: Part 1: A cross-sectional study aims to investigate the influence of fatigue on the MI ability in PD compared to healthy controls Part 2: A randomized controlled trial compare the effect of fNIRS-based NFB-MI on balance and gait performance versus MI and MT group in people with PD.
Who Masked: Outcomes Assessor
Masking Description: Assessor will be blinded to the allocation until the last assessment (4-week follow-up).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Neurofeedback combined with MI (NFB-MI) (Experimental): Participants in both NFB-MI and MI groups will receive a total of 12 sessions of training in 4 weeks. NFB-MI group will receive fNIRS-based neurofeedback during MI training in lab. Prior to each NFB-MI session, participants will watch a video of a person executing balance tasks and walking in different environments. The explicit instruction will be given by the researcher. Each MI training session (consisting of 5 trials for balance and walking tasks) includes 45 seconds of imagery tasks followed by 15 seconds of rest, repeated twice. The training will take approximately 20 minutes. Visual feedback with a thermometer based on the changes of HbO concentration will be displayed on the screen during NFB-MI training.
  In each training session, actual balance and gait tasks will be practiced for 20 min. The difficulty of the tasks will be modified individually for each participant.
  Interventions: Other: fNIRS-based neurofeedback with motor imagery; Other: Motor training
- Motor imagery (Active Comparator): Participants in both NFB-MI and MI groups will receive a total of 12 sessions of training in 4 weeks. MI group will practice kinesthetic MI under supervision in lab setting. Participants will watch a video of a person executing balance tasks and walking in different environments before MI training. The explicit instruction will be given by the researcher. Each MI training session (consisting of 5 trials for balance and walking tasks) includes 45 seconds of imagery tasks followed by 15 seconds of rest, repeated twice. The training will take approximately 20 minutes.
  In each training session, actual balance and gait tasks will be practiced for 20 min after MI training. The difficulty of the tasks will be modified individually for each participant. The researcher will ensure the safety of executing each task during lab visit.
  Interventions: Other: Kinesthetic motor imagery; Other: Motor training
- Motor training (Active Comparator): The tasks for balance and gait training are similar to those during the MI training. The balance and gait training will be practiced for 20 min in MI and NFB-MI groups, and will be practiced for 40 min in MT group. The difficulty of the tasks will be modified individually for each participant. The researcher will ensure the safety.
  Interventions: Other: Motor training

INTERVENTIONS:
Other: fNIRS-based neurofeedback with motor imagery — A multichannel wearable fNIRS (NIRSport2, NIRx Medical Technologies LLC, Glen Head, NY, USA) will be used to detect the cortical activity in SMA. The HbO concentration will be processed and displayed as a visual feedback during MI training.
  Arms: Neurofeedback combined with MI (NFB-MI)
Other: Kinesthetic motor imagery — Prior to each task, participants will watch a video of a person executing balance tasks and walking tasks. The balance tasks will include static and dynamic standing tasks such as sit-to-stand, tandem stance, standing on a balance board, reaching out to different directions and single leg stance. The walking tasks consists of tandem walking, crossing obstacles, sideward walking, backward walking, and turning. The participants will be asked to kinesthetically imagine movements in the first-person perspective, and the researcher will give the explicit instruction encouraging them to focus on the feeling (i.e. tactile, proprioceptive and kinesthetic sensations). Each MI session consists of 10-min of balance tasks and 10-min of walking tasks.
  Arms: Motor imagery
Other: Motor training — The tasks for balance and gait training are similar to those during the MI training. The difficulty of the tasks will be modified individually for each participant. The researcher will ensure the safety.

SUMMARY:
A cross-sectional study (part 1) aims to investigate the influence of fatigue on the MI ability in PD compared to healthy controls. A randomized controlled trial (part 2) aims to compare the effect of fNIRS-based NFB-MI on balance and gait performance versus MI only in people with PD.

DETAILED DESCRIPTION:
To fulfill out study purposes, a cross-sectional study (Part I) and an interventional randomized controlled trial (Part II) are designed. In Part I, people with PD and the age-matched healthy controls will be recruited and perform imagery and actual walking tasks. The level of general fatigue will be measured by Traditional Chinese version of Multidimensional Fatigue Inventory (MFI-TC) in people with PD. The level of concurrent fatigue will be induced by 30-minute cognitive tasks consisting of A-X continuous performance test, 2 back and mental rotation test and will be assessed by Brunel Mood Scale (BRUMS-C) in people with PD. Independent t test will be used to compare the MI ability between PD group and healthy control group. The Pearson's correlation coefficient will be used to examine the relationships between general fatigue level (MFI) and MI ability and between concurrent fatigue level (BRUMS) and MI ability in people with PD. In Part II, people with PD will be randomly allocated to either NFB-MI, MI or MT group. Every participant will receive 12 sessions of training in four weeks. NFB-MI and MI training will consist of 20-min MI with or without neurofeedback respectively followed by 20-min of balance and gait training. In the MT group, participants will receive 40-min of balance and gait training. Outcome measures, including Mini Balance Evaluation Systems Test (Mini-BEST), Timed up-and-go test (TUG), gait performance, will be assessed at pre-, post-test, and follow-up. MI ability and fatigue will be assessed at pre-, mid-and post-test. A two-way analysis of variance (ANOVA) with repeated measure will be used to determine the time by group interaction for all the outcomes. Post hoc test with Bonferroni correction will be applied for significant interaction. Significant level for part I and part II will be set at p < 0.05.

ELIGIBILITY:
Part 1

Additional Inclusion Criteria for PD:

1. diagnosis of idiopathic PD by neurologist with Hoehn and Yahr stage < 4;
2. stable medical condition;
3. capability of walking independently without walking devices.

Exclusion Criteria:

1. cognitive impairment indicated by MMSE score < 24;
2. motor imagery ability indicated by KVIQ score < 25;
3. unable recognize 26 letters in the English alphabet
4. history of diseases or conditions known to interfere with participating this study (e.g. epilepsy, metal implants in the brain, or deep brain stimulation);
5. diagnosis of any other neurological disease or psychiatric disorder (e.g. stroke, anxiety disorder, or depression);
6. using central nervous system medications other than for PD, e.g. antiepileptic drugs in recent 3 months.

Part 2

Inclusion Criteria:

1. aged 40-85 y/o;
2. diagnosis of idiopathic PD by neurologist with Hoehn and Yahr stage < 4;
3. stable medical condition;
4. capability of walking independently for 10 minutes, which is the time needed for imagery walking training in order to eliminate the possible influence of physical fatigue.

Exclusion Criteria:

1. cognitive impairment indicated by MMSE score < 24;
2. history of diseases or conditions known to interfere with participating this study (e.g. epilepsy, metal implants in the brain, or deep brain stimulation);
3. diagnosis of any other neurological disease or psychiatric disorder (e.g. stroke, anxiety disorder, or depression);
4. using central nervous system medications other than for PD, e.g. antiepileptic drugs in recent 3 months.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 93 (Estimated)
Dates: Start 2025-03-19 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Self-perceived fatigue for general fatigue level | Part 1 cross-sectional assessment (day 1 of the study)
  Traditional Chinese version of Multidimensional Fatigue Inventory (MFI-TC) will be used to measure subjective perception of fatigue. MFI-TC is a 20-item self-report scale evaluating different dimensions of fatigue (general fatigue/physical fatigue, reduced activity, reduced motivation and mental fatigue). Each item is scored on a 1 (strongly agree) to 5 (strongly disagree) scale to assess how well the statement describe the participant's experience of fatigue. Ten positively phrased items (item 2, 5, 9, 10, 13, 14, 16, 17, 18, 19) were reverse-scored before adding up scores. The total score obtained simply by adding 20-item scores together (i.e., 20-100), with higher scores indicating more fatigue.
Motor imagery ability | Part 1 cross-sectional assessment (day 1 of the study and day 8 for second assessment)
  The walking tasks during motor imagery: walkways of 5 m in length, and 35 cm in width. Participants will be asked to stand upright at the starting line, and then perform imagery walking (IW) and actual walking (AW) task in a total of 2 sessions in the following sequence: IW- walkway (35cm), and AW- walkway. Each session contains three repeated trials of walking over 5 m walkways. The MI ability will be indicated by the index of performance (IP) calculated by [(AW - IW/ AW) * 100]. IP closer to zero indicates better MI ability.
Kinesthetic and visual imagery ability | Part 1 cross-sectional assessment (day 1 of the study and day 8 for second assessment)
  Kinesthetic and visual imagery questionnaire-short version (KVIQ-10) will be used to assess kinesthetic and visual imagery ability. 5 movement will be demonstrated by the assessor and mimicked by the participant. The participant will be asked to visually and kinesthetically imagine the movement without doing the movement. The clarity of the image (visual subscale) and the intensity of the sensations (kinesthetic subscale) will be scored on a five point ordinal scale. The total scores ranged from 10 to 50, and higher scores indicate better ability on kinesthetic and visual imagery.
Self-perceived fatigue for concurrent fatigue level | Part 1 cross-sectional assessment (day 8 of the study)
  Chinese version of the Brunel Mood Scale (BRUMS-C) will be used to measure subjective perception of fatigue. Fatigue is a subscale of BRUMS-C consisted with 4-item. Participants indicated whether they have felt on a five-point Likert scale (0 = not at all,1 = a little, 2 = moderately, 3 = quite a bit, 4 = extremely) using the "How do you feel right now?" response timeframe. The total score obtained simply by adding 4-item scores together (i.e., 0-16), with higher scores indicating more fatigue.
Change of Mini Balance Evaluation Systems Test (Mini-BEST) from pre-test to post-test | Part 2 pre-test, post-test (4 weeks)
  Mini-BEST is used to measure dynamic balance ability in four domains: anticipatory postural adjustment, reactive postural adjustments, sensory integration and dynamic gait. Mini-BEST consists of 14 items scored on a 0-2 scale, with 2 items assess right and left sides. The total scores will be 0-32, and higher scores indicate better balance ability. The scores at pre-test subtracting from the scores at post-test will be presented.
Change of Mini Balance Evaluation Systems Test (Mini-BEST) from pre-test to follow-up | Part 2 pre-test and 4-week follow-up assessment (8 weeks)
  Mini-BEST is used to measure dynamic balance ability in four domains: anticipatory postural adjustment, reactive postural adjustments, sensory integration and dynamic gait. Mini-BEST consists of 14 items scored on a 0-2 scale, with 2 items assess right and left sides. The total scores will be 0-32, and higher scores indicate better balance ability.The scores at pre-test subtracting from the scores at follow-up will be presented.
Change of Timed up-and-go test (TUG) from pre-test to post-test | Part 2 pre-test and post-test (4 weeks)
  Functional mobility will be indicated by TUG. Participants will be asked to stand up from a chair, walk at comfortable speed for 3 m, turn around and sit back on the chair. The completing duration will be measured, and the mean value across 3 trials of TUG will be documented as the final performance. The shorter completing duration indicates better mobility function. The duration at pre-test subtracting from the duration at post-test will be presented.
Change of Timed up-and-go test (TUG) from pre-test to follow-up | Part 2 pre-test and 4-week follow-up assessment (8 weeks)
  Functional mobility will be indicated by TUG. Participants will be asked to stand up from a chair, walk at comfortable speed for 3 m, turn around and sit back on the chair. The completing duration will be measured, and the mean value across 3 trials of TUG will be documented as the final performance. The shorter completing duration indicates better mobility function. The duration at pre-test subtracting from the duration at follow-up will be presented.
Change of gait performance from pre-test to post-test | Part 2 pre-test and post-test (4 weeks)
  The gait parameters will be measured by a GAITRite system (CIR system, Inc., Havertown, Pennsylvania). The GAITRite system is a 4.57 m long, 0.9 m wide straight walkway containing pressure-sensitive sensors in a 3.66 m by 0.61 m area. The participants will be instructed to walk along the walkway at their comfortable speed for 3 times. The values at pre-test subtracting from the values at post-test will be presented.
Change of gait performance from pre-test to follow-up | Part 2 pre-test and 4-week follow-up assessment (8 weeks)
  The gait parameters will be measured by a GAITRite system (CIR system, Inc., Havertown, Pennsylvania). The GAITRite system is a 4.57 m long, 0.9 m wide straight walkway containing pressure-sensitive sensors in a 3.66 m by 0.61 m area. The participants will be instructed to walk along the walkway at their comfortable speed for 3 times. The values at pre-test subtracting from the values at follow-up will be presented.

SECONDARY OUTCOMES:
Change of self-perceived fatigue from pre-test to mid-test | Part 2 pre-test and mid-test (2 weeks)
  Traditional Chinese version of Multidimensional Fatigue Inventory (MFI-TC) will be used to measure subjective perception of fatigue. MFI-TC is a 20-item self-report scale evaluating different dimensions of fatigue (general fatigue/physical fatigue, reduced activity, reduced motivation and mental fatigue). Each item is scored on a 1 (strongly agree) to 5 (strongly disagree) scale to assess how well the statement describe the participant's experience of fatigue. Ten positively phrased items (item 2, 5, 9, 10, 13, 14, 16, 17, 18, 19) were reverse-scored before adding up scores. The total score obtained simply by adding 20-item scores together (i.e., 20-100), with higher scores indicating more fatigue. The scores at pre-test subtracting from the scores at mid-test will be presented.
Change of self-perceived fatigue from pre-test to post-test | Part 2 pre-test and post-test (4 weeks)
  Traditional Chinese version of Multidimensional Fatigue Inventory (MFI-TC) will be used to measure subjective perception of fatigue. MFI-TC is a 20-item self-report scale evaluating different dimensions of fatigue (general fatigue/physical fatigue, reduced activity, reduced motivation and mental fatigue). Each item is scored on a 1 (strongly agree) to 5 (strongly disagree) scale to assess how well the statement describe the participant's experience of fatigue. Ten positively phrased items (item 2, 5, 9, 10, 13, 14, 16, 17, 18, 19) were reverse-scored before adding up scores. The total score obtained simply by adding 20-item scores together (i.e., 20-100), with higher scores indicating more fatigue. The scores at pre-test subtracting from the scores at post-test will be presented.
Change of motor imagery ability from pre-test to mid-test | Part 2 pre-test and mid-test (2 weeks)
  There are two conditions for walking tasks during motor imagery: wide and narrow walkways of 15 m in length, and respectively 2 m and 35 cm in width. participants will be asked to stand upright at the starting line, and then perform imagery walking (IW) and actual walking (AW) task in a total of four sessions in the following sequence: IW-wide walkway (2m), AW-wide walkway, IW-narrow walkway (35cm), and AW-narrow walkway. Each session contains three repeated trials of walking over 15 m wide or narrow walkways. The MI ability will be indicated by the index of performance (IP) calculated by [(AW - IW/ AW) * 100]. IP closer to zero indicates better MI ability. The scores at pre-test subtracting from the scores at mid-test will be presented.
Change of motor imagery ability from pre-test to post-test | Part 2 pre-test and post-test (4 weeks)
  There are two conditions for walking tasks during motor imagery: wide and narrow walkways of 15 m in length, and respectively 2 m and 35 cm in width. participants will be asked to stand upright at the starting line, and then perform imagery walking (IW) and actual walking (AW) task in a total of four sessions in the following sequence: IW-wide walkway (2m), AW-wide walkway, IW-narrow walkway (35cm), and AW-narrow walkway. Each session contains three repeated trials of walking over 15 m wide or narrow walkways. The MI ability will be indicated by the index of performance (IP) calculated by [(AW - IW/ AW) * 100]. IP closer to zero indicates better MI ability. The scores at pre-test subtracting from the scores at post-test will be presented.
Change of kinesthetic and visual imagery ability from pre-test to mid-test | Part 2 pre-test and mid-test (2 weeks)
  Kinesthetic and visual imagery questionnaire-short version (KVIQ-10) will be used to assess kinesthetic and visual imagery ability. 5 movement will be demonstrated by the assessor and mimicked by the participant. The participant will be asked to visually and kinesthetically imagine the movement without doing the movement. The clarity of the image (visual subscale) and the intensity of the sensations (kinesthetic subscale) will be scored on a five point ordinal scale. The total scores ranged from 10 to 50, and higher scores indicate better ability on kinesthetic and visual imagery. The scores at pre-test subtracting from the scores at mid-test will be presented.
Change of kinesthetic and visual imagery ability from pre-test to post-test | Part 2 pre-test and post-test (4 weeks)
  Kinesthetic and visual imagery questionnaire-short version (KVIQ-10) will be used to assess kinesthetic and visual imagery ability. 5 movement will be demonstrated by the assessor and mimicked by the participant. The participant will be asked to visually and kinesthetically imagine the movement without doing the movement. The clarity of the image (visual subscale) and the intensity of the sensations (kinesthetic subscale) will be scored on a five point ordinal scale. The total scores ranged from 10 to 50, and higher scores indicate better ability on kinesthetic and visual imagery. The scores at pre-test subtracting from the scores at post-test will be presented.

CONTACTS AND LOCATIONS:
Overall Officials: Ray-Yau Wang, Principal Investigator — National Yang Ming Chiao Tung University
Locations (1):
- National Yang Ming Chiao Tung University, Taipei, None Selected, Taiwan